CLINICAL TRIAL: NCT01955694
Title: A Randomized, Double-blind, Double-dummy, Multi-center Study to Assess Safety and Efficacy of BAY94-8862 in Japanese Subjects With Emergency Presentation at the Hospital Because of Worsening Chronic Heart Failure With Left Ventricular Systolic Dysfunction and Either Type 2 Diabetes Mellitus With or Without Chronic Kidney Disease or Moderate Chronic Kidney Disease Alone Versus Eplerenone
Brief Title: Phase IIb Safety and Efficacy Study of BAY94-8862 in Subjects With Worsening Chronic Heart Failure and Left Ventricular Systolic Dysfunction and Either Type 2 Diabetes Mellitus With or Without Chronic Kidney Disease or Moderate Chronic Kidney Disease Alone
Acronym: ARTS-HF Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16815
Record Dates: First submitted 2013-09-30; First posted 2013-10-07 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: BAY94-8862; MR antagonist; Heart failure; Japanese patients
MeSH Terms: conditions — Heart Failure | interventions — finerenone; Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- BAY94-8862 (2.5 mg) (Experimental): 2.5 mg BAY94-8862 tablet and placebo capsule once daily in the morning, with possible up-titration to 5 mg once daily at Visit 6 (Day 30), and sham up-titration at Visit 8 (Day 60), based on the value of blood potassium
  Interventions: Drug: BAY94-8862; Drug: Placebo
- BAY94-8862 (5 mg) (Experimental): 5 mg BAY94-8862 tablet and placebo capsule once daily in the morning, with possible up-titration to 10 mg once daily at Visit 6 (Day 30), and sham up-titration at Visit 8 (Day 60), based on the value of blood potassium
  Interventions: Drug: BAY94-8862; Drug: Placebo
- Eplerenone (Active Comparator): 25 mg eplerenone every other day, i.e. one 25 mg eplerenone capsule on Day 1, Day 3, Day 5, etc. in the morning, 1 placebo capsule on Day 2, Day 4, Day 6, etc. in the morning, and 1 placebo tablet once daily in the morning, with possible up-titration to 25 mg eplerenone once daily at Visit 6 (Day 30), i.e. one 25 mg eplerenone capsule once daily in the morning and 1 placebo tablet once daily in the morning, and a possible up-titration to 25 mg once daily [if not performed at Visit 6 (Day 30)] or to 50 mg once daily [if up-titrated to 25 mg once daily at Visit 6 (Day 30)] at Visit 8 (Day 60), based on the value of blood potassium
  Interventions: Drug: Eplerenone; Drug: Placebo
- BAY94-8862 (7.5 mg) (Experimental): 7.5 mg BAY94-8862 tablet and placebo capsule once daily in the morning, with possible up-titration to 15 mg once daily at Visit 6 (Day 30), and sham up-titration at Visit 8 (Day 60), based on the value of blood potassium Note: This treatment group may be introduced into the study or not after safety and tolerability of these doses has been assessed by an independent Data Monitoring Committee (DMC) (1st dose recommendation DMC meeting).
  Interventions: Drug: BAY94-8862; Drug: Placebo
- BAY94-8862 (10 mg) (Experimental): 10 mg BAY94-8862 tablet and placebo capsule once daily in the morning, with possible up-titration to 20 mg once daily at Visit 6 (Day 30), and sham up-titration at Visit 8 (Day 60), based on the value of blood potassium Note: Only in case the above mentioned additional treatment arm (BAY94-8862, 7.5 mg) has been added, a second dose decision meeting of the DMC will take place, Again safety and tolerability of all doses will be assessed by an independent DMC (2nd dose recommendation DMC meeting). Based on this data, none or up to two treatment groups (BAY94-8862, 10 mg and BAY94-8862,15 mg) may be introduced into the study.
  Interventions: Drug: BAY94-8862; Drug: Placebo
- BAY94-8862 (15 mg) (Experimental): 15 mg BAY94-8862 tablet and placebo capsule once daily in the morning, with possible up-titration to 20 mg once daily at Visit 6 (Day 30), and sham up-titration at Visit 8 (Day 60), based on the value of blood potassium Note: Only in case the above mentioned additional treatment arm (BAY94-8862, 7.5 mg) has been added, a second dose decision meeting of the DMC will take place, Again safety and tolerability of all doses will be assessed by an independent DMC (2nd dose recommendation DMC meeting). Based on this data, none or up to two treatment groups (BAY94-8862, 10 mg and BAY94-8862,15 mg) may be introduced into the study.
  Interventions: Drug: BAY94-8862; Drug: Placebo

INTERVENTIONS:
Drug: BAY94-8862 — 2.5 mg, 5 mg, 7.5 mg, 10 mg, 15 mg, and 20 mg of BAY94-8862 tablets
  Arms: BAY94-8862 (10 mg); BAY94-8862 (15 mg); BAY94-8862 (2.5 mg); BAY94-8862 (5 mg); BAY94-8862 (7.5 mg)
Drug: Eplerenone — INSPRA 25 and 50 mg tablets (MAH: Pfizer) will be used for eplerenone 25 and 50 mg tablets
  Arms: Eplerenone
Drug: Placebo — matching placebo

SUMMARY:
This study will be conducted in subjects with clinical diagnosis of worsening chronic heart failure and either type 2 diabetes mellitus (DM) with or without chronic kidney disease (CKD) or moderate CKD alone treated with evidence-based therapy for heart failure (HF) for at least 3 months prior to emergency presentation to hospital using a multi-center, randomized, adaptive, double-blind, double-dummy, comparator-controlled, parallel-group design.

Primary objective of the study is to investigate efficacy [percentage of subjects with a relative decrease in N-terminal prohormone B-type natriuretic peptide (NT-proBNP) of more than 30% from baseline to Visit 10 (Day 90)] and safety of different oral doses of BAY94-8862 given once daily.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with worsening chronic heart failure requiring emergency presentation to hospital and treatment with intravenous (IV) diuretics at hospital
* Subjects with either type 2 DM or moderate CKD

Exclusion Criteria:

* Acute de-novo heart failure or acute inflammatory heart disease, e.g. acute myocarditis
* Acute coronary syndrome (ACS) (elevated cardiac troponins which are not caused by an ACS are not an exclusion criterion) in the last 30 days prior to the screening visit
* Cardiogenic shock
* Valvular heart disease requiring surgical intervention during the course of the study
* Subjects with left ventricular assistance device or waiting for heart transplantation
* Stroke or transient ischemic cerebral attack in the last 3 months prior to the screening visit
* Addison's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2015-01-23 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with a relative decrease in N-terminal prohormone B-type natriuretic peptide of more than 30% from baseline to Visit 10 | From baseline to 90 days

SECONDARY OUTCOMES:
Change in serum potassium | From baseline to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (26):
- Japan (26):
  - Seto, Aichi-ken
  - Toyota, Aichi-ken
  - Funabashi, Chiba
  - Kamogawa, Chiba
  - Matsuyama, Ehime
  - Chikushino-shi, Fukuoka
  - Amagasaki, Hyōgo
  - Kobe, Hyōgo
  - Higashiibaraki, Ibaraki
  - Hiratsuka, Kanagawa
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Uji, Kyoto
  - Sendai, Miyagi
  - Naha, Okinawa
  - Urasoe, Okinawa
  - Sayama, Saitama
  - Kusatsu, Shiga
  - Shinjuku-ku, Tokyo
  - Kofu, Yamanashi
  - Fukuoka
  - Kagoshima
  - Kyoto
  - Okayama
  - Osaka
  - Shizuoka

REFERENCES:
- [Result] Sato N, Ajioka M, Yamada T, Kato M, Myoishi M, Yamada T, Kim SY, Nowack C, Kolkhof P, Shiga T; ARTS-HF Japan study group. A Randomized Controlled Study of Finerenone vs. Eplerenone in Japanese Patients With Worsening Chronic Heart Failure and Diabetes and/or Chronic Kidney Disease. Circ J. 2016 Apr 25;80(5):1113-22. doi: 10.1253/circj.CJ-16-0122. Epub 2016 Apr 14. PMID 27074824
- See also: Click here to find results for studies related to Bayer Healthcare products. — http://clinicaltrials.bayer.com/